CLINICAL TRIAL: NCT02822651
Title: SCOPYD Study: Development of a Predictive Clinical Score of Hypovitaminosis D
Brief Title: Hypovitaminosis D Prediction Score
Acronym: SCOPYD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL15_0078
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Vitamin D Status
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D status (Experimental): The 2500 subjects included in this unique arm will complete a self-administered questionnaire and will have a blood sampling to measure vitamin D blood concentration.
  Interventions: Biological: Blood sampling; Other: self-administered questionnaire

INTERVENTIONS:
Biological: Blood sampling — Patients will have a blood sampling at inclusion to measure vitamin D blood concentration.
Other: self-administered questionnaire — Patients will fill a self-administered questionnaire the day of inclusion

SUMMARY:
Vitamin D has effects on many tissues, and hypovitaminosis D is frequent. In a French survey conducted among 1587 adults, vitamin D insufficiency (<30ng/ml) has been reported in 80% of subjects, including 43% with moderate deficiency (<20ng/ml) and 5% with severe deficiency (<10ng/ml).

Because of the possible consequences of hypovitaminosis D (osteomalacia in adults…), the number of vitamin D determination has increased ten-fold since 2005 in France, reaching 4.5 million € in 2011, and with it the costs for health insurance. However, there is currently no consensus on the strategy for detection, diagnosis and treatment of hypovitaminosis D.

We propose to develop a predictive clinical score of hypovitaminosis D based on the accurate assessment of solar exposure, vitamin D intakes and hypovitaminosis D risk factors collected through a self-administered questionnaire.

ELIGIBILITY:
Inclusion Criteria:

- Men and women aged 18 to 70 years old

Exclusion Criteria:

* Participation in a study related to vitamin D
* Taking at least 80 000 IU vitamin D in the last 3 months as a single dose
* Pregnancy or breast-feeding
* Renal failure : severe renal impairment, dialysis, having kidney transplant
* Known hepatic impairment
* Gastrointestinal disorders: Celiac disease, Crohn's disease, ulcerative colitis, bariatric surgery, gastrointestinal surgery with stoma
* Known primary hypo/hyperparathyroidism
* Bone cancer/metastases current or in the last 2 years
* Treatment with antiepileptics
* Long-term treatment with glucocorticoids (> 3 months)
* Treatment with antiretroviral
* Legal incapacity or limited legal capacity
* Non-recipient of French Social Security

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2592 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
25 (OH) vitamin D blood concentration | The day of inclusion
  Vitamin D determination will be carried out for each center in a single laboratory by chemiluminescence technique.
  Vitamin D determination is the gold standard for the development and validation phases of the score. It will define the variables of the self-administered questionnaire to be included in the final score (development phase) and be the gold standard in the evaluation of the performance score (validation phase). The blood sample will be collected after the completion of the questionnaire, on the same day.

SECONDARY OUTCOMES:
Vitamin D concentration level | The day of inclusion
  The ability of the score to classify adults in one of these three categories:
  * Category 1 : Vitamin D sufficiency (≥30 ng/ml)
  * Category 2 : Hypovitaminosis D between 30 and 10 ng/ml
    * Vitamin D insufficiency (<30 ng/ml)
    * Vitamin D deficiency (<20 ng/ml)
  * Category 3 : Severe deficiency (<10 ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie SCHOTT-PETHELAZ, MD, PhD, Principal Investigator — Hospices Civils de Lyon - Pôle d'Information Médicale et d'Evaluation de la Recherche
Locations (1):
- Hospices Civils de Lyon - Pôle IMER, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Viprey M, Merle B, Riche B, Freyssenge J, Rippert P, Chakir MA, Thomas T, Malochet-Guinamand S, Cortet B, Breuil V, Chapurlat R, Lafage Proust MH, Carlier MC, Fassier JB, Haesebaert J, Caillet P, Rabilloud M, Schott AM. Development and Validation of a Predictive Model of Hypovitaminosis D in General Adult Population: SCOPYD Study. Nutrients. 2021 Jul 23;13(8):2526. doi: 10.3390/nu13082526. PMID 34444687